CLINICAL TRIAL: NCT04417907
Title: Effects of Titration Rate on Cognitive and Behavioral Side Effects of Perampanel
Brief Title: Perampanel Titration and Cognitive Effects
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study sponsor no longer provided funding.
Sponsor: Kimford Jay Meador (Other)
Collaborators: Eisai Inc. (Industry)
Responsible Party: Sponsor-Investigator, Kimford Jay Meador, Professor of Neurology and Neurological Sciences, Stanford University
Organization: Stanford University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 54358
Record Dates: First submitted 2020-06-02; First posted 2020-06-05 (Actual); Results first posted 2024-06-06 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-05

CONDITIONS: Epilepsy
Keywords: Perampanel; Cognition
MeSH Terms: conditions — Epilepsy | interventions — perampanel

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): Participants will take 2mg placebo PO QD for six weeks.
  Interventions: Drug: Placebo
- PER 1 Week Titration (Experimental): Participants will take 2mg perampanel PO QD for one week, followed by 4mg perampanel PO QD for five weeks.
  Interventions: Drug: Perampanel 1 week titration
- PER 2 Week Titration (Experimental): Participants will take 2mg perampanel PO QD for two weeks, followed by 4mg perampanel PO QD for four weeks.
  Interventions: Drug: Perampanel 2 week titration
- PER 4 mg (Experimental): Participants will take 4mg perampanel PO QD for six weeks
  Interventions: Drug: Perampanel 4mg

INTERVENTIONS:
Drug: Perampanel 1 week titration — Healthy adults will take 2mg perampanel PO QD for one week followed 4mg perampanel PO QD for five weeks.
  Other Names: Fycompa
  Arms: PER 1 Week Titration
Drug: Perampanel 2 week titration — Healthy adults will take 2mg perampanel PO QD for two weeks followed 4mg perampanel PO QD for four weeks.
  Other Names: Fycompa
  Arms: PER 2 Week Titration
Drug: Perampanel 4mg — Healthy adults will take 4mg perampanel PO QD for six weeks
  Other Names: Fycompa
  Arms: PER 4 mg
Drug: Placebo — Healthy adults will take 2mg placebo PO QD for six weeks
  Arms: Placebo

SUMMARY:
The objective of this study is to determine whether there are any differences in the cognitive abilities and/or behavioral response of normal healthy volunteers across different titration rates of perampanel.

DETAILED DESCRIPTION:
This is a randomized, double-blind, parallel group design across different titration rates of perampanel in healthy volunteers. The study consists of 8 visits, 4 of which will occur at the participant's home, over a 7-week period. One hundred and three (103) normal healthy subjects will be treated with perampanel (PER) at one of four different titration rates: (1) 2mg/day PER for one week followed by 4mg/day PER for five weeks, (2) 2mg/day PER for two weeks followed by 4mg/day PER for four weeks, (3) 4mg/day PER for six weeks, or (4) placebo (0mg/day PER) for six weeks. Cognitive and behavioral function testing along with safety testing will be conducted at screening, pretreatment baseline, the end of each week during the titration and maintenance period.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults between the ages of 18 and 55 years
2. Male or female (using approved birth control methods)
3. Informed consent obtained

Exclusion Criteria:

1. Presence of clinically significant cardiovascular, endocrine, hematopoietic, hepatic, neurologic, psychiatric, or renal disease.
2. Presence or history of drug or alcohol abuse or positive urine drug test at screening.
3. The use of concomitant medications, which are known to affect perampanel or the use of any concomitant medications that may alter cognitive function (see Section VIII.F for a partial list).
4. Prior adverse reaction to or prior hypersensitivity to perampanel.
5. Prior participation in studies involving perampanel.
6. Subjects who have received any investigational drug within the previous thirty days.
7. Subjects with IQ < 80 as determined by the Peabody Picture Vocabulary Test after enrollment.
8. Positive pregnancy test. Women of childbearing potential will be required to use approved birth control methods during the study.
9. Presence of lifetime history of suicide attempt (including an active attempt, interrupted attempt, or aborted attempt), or has suicidal ideation in the past 6 months as indicated by a positive response ('Yes') to either Question 4 or Question 5 of the C-SSRS at Screening.
10. Invalid results on computerized cognitive tests at screening as indicated by a 'No' on any of the validity indicators generated in the CNS Vital Signs report.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2021-10-20 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kimford Meador, MD, Principal Investigator — Stanford University
Locations (3):
- United States (3):
  - Stanford University, Palo Alto, California
  - Northwestern University, Chicago, Illinois
  - New York University, New York, New York

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants take 2mg placebo PO QD for six weeks.
- PER 1 Week Titration: Participants take 2mg perampanel PO QD for one week and 4mg perampanel PO QD for five weeks.
- PER 2 Week Titration: Participants take 2mg perampanel PO QD for two weeks and 4mg perampanel PO QD for four weeks.
- PER 4 mg: Participants take 4mg perampanel PO QD for six weeks
Period: Overall Study
Arm/Group | Placebo | PER 1 Week Titration | PER 2 Week Titration | PER 4 mg
Started | 4 | 7 | 7 | 11
Completed | 2 | 3 | 6 | 8
Not Completed | 2 | 4 | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | PER 1 Week Titration | PER 2 Week Titration | PER 4 mg | Total
Number analyzed (Participants) | 4 | 7 | 7 | 11 | 29
Age, Continuous [Mean (Standard Deviation); unit: Years] | 44.8 (10.3) | 34.7 (10.3) | 30.3 (8.9) | 39.7 (12.8) | 36.9 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 3 | 5 | 16
  Male | 1 | 2 | 4 | 6 | 13
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 1 | 2 | 2 | 5
  Black/African American | 1 | 0 | 1 | 2 | 4
  Hispanic/Latino | 1 | 2 | 2 | 0 | 5
  White/Caucasian | 2 | 4 | 1 | 6 | 13
  Other | 0 | 0 | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 4 | 7 | 7 | 11 | 29
Education Level [Mean (Standard Deviation); unit: Years] — Education level was assessed by asking participants their highest level of education. Participants' responses was then converted to the number of years this level of education corresponds to.
  Years | 16 (1.6) | 17 (1.9) | 16 (1.2) | 15.7 (2.2) | 16.1 (1.8)
IQ Estimate [Mean (Standard Deviation); unit: units on a scale] — IQ estimate is the Peabody Picture Vocabulary Test, 4th ed. (PPVT-4). The overall standard score is reported. Ranges are 40 to 160. Higher scores indicate better performance.
  units on a scale | 99 (7.1) | 102.3 (6.7) | 97.1 (11) | 102.9 (7.4) | 100.8 (8.2)

OUTCOME MEASURES:

1. Primary Outcome: Overall Neuropsychological Composite Z-score as a Measure of Direct Comparison of the 4 Titration Conditions Across 6 Weeks of Treatment.
Description: Z score of cognitive tests (selected performance measures from the computerized cognitive test battery) and questionnaires (AEP, POMS, QOLIE-cognitive questions) at the end of each week of drug treatment for each titration arm, controlling for baseline measures collected prior to treatment. Various measures were combined collectively (averaged) to compute an overall Z-score for each group at each time point. These included: 1) Executive Function Score of computerized test battery; 2) Processing Speed Score of computerized test battery; 3) AEP total score; 4) POMS total and domain scores; 5) Three cognitive components of the QOLIE-31 (attention, memory, language). The Z-score indicates the number of standard deviations away from a reference population. A Z-score of 0 is equal to the mean. Negative numbers indicate poorer performance compared to the mean and positive numbers represent higher performance compared to the mean.
Time Frame: At the end of each week of treatment for 6 weeks.
Population: Participants who completed the protocol are included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | PER 1 Week Titration | PER 2 Week Titration | PER 4 mg
Number analyzed (Participants) | 2 | 3 | 6 | 8
score on a scale
  Week 1 | -.41 (1.00) | -.07 (.55) | .05 (.28) | .32 (.33)
  Week 2 | -.25 (.90) | -.01 (.44) | -.15 (.26) | .15 (.27)
  Week 3 | -.14 (.71) | -.03 (.36) | .02 (.34) | .10 (.34)
  Week 4 | -.32 (.81) | -.06 (.40) | .09 (.49) | .23 (.33)
  Week 5 | -.34 (.85) | -.11 (.53) | -.03 (.35) | .37 (.41)
  Week 6 | -.28 (.87) | -.03 (.45) | -.11 (.35) | .21 (.48)

2. Primary Outcome: Composite Z-score of Objective Measures as a Measure of Direct Comparison of the 4 Titration Conditions Across 6 Weeks of Treatment.
Description: Z score of objective cognitive tests (selected performance measures from the computerized cognitive test battery) at the end of each week of drug treatment for each titration arm, controlling for baseline measures collected prior to treatment. The Z-score indicates the number of standard deviations away from a reference population. A Z-score of 0 is equal to the mean. Negative numbers indicate poorer performance compared to the mean and positive numbers represent higher performance compared to the mean.
Time Frame: At the end of each week of treatment for 6 weeks.
Population: Participants who completed the protocol are included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | PER 1 Week Titration | PER 2 Week Titration | PER 4 mg
Number analyzed (Participants) | 2 | 3 | 6 | 8
score on a scale
  Week 1 | -.69 (.52) | .61 (.21) | .04 (.38) | .11 (.23)
  Week 2 | .26 (.03) | .44 (.20) | -.05 (.02) | .11 (.40)
  Week 3 | .04 (.30) | .24 (.30) | .05 (.12) | .11 (.11)
  Week 4 | .51 (.15) | .28 (.23) | -.17 (.38) | .27 (.31)
  Week 5 | .06 (.19) | .33 (.02) | -.15 (.01) | .07 (.08)
  Week 6 | .28 (.25) | .11 (.38) | -.21 (.34) | -.06 (.37)

3. Primary Outcome: Composite Z-score of Subjective Measures as a Measure of Direct Comparison of the 4 Titration Conditions Across 6 Weeks of Treatment.
Description: Z score of subjective questionnaires (AEP, POMS, QOLIE-cognitive questions at the end of each week of drug treatment for each titration arm, controlling for baseline measures collected prior to treatment. Various measures were combined collectively (averaged) to compute an overall Z-score for each group at each time point. These included: 1) AEP total score; 2) POMS total and domain scores; 3) Three cognitive components of the QOLIE-31 (attention, memory, language). The Z-score indicates the number of standard deviations away from a reference population. A Z-score of 0 is equal to the mean. Negative numbers indicate poorer performance compared to the mean and positive numbers represent higher performance compared to the mean.
Time Frame: At the end of each week of treatment for 6 weeks.
Population: Participants who completed the protocol are included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | PER 1 Week Titration | PER 2 Week Titration | PER 4 mg
Number analyzed (Participants) | 2 | 3 | 6 | 8
score on a scale
  Week 1 | -.36 (1.08) | -.20 (.50) | .05 (.28) | .36 (.34)
  Week 2 | -.35 (.96) | -.09 (.43) | -.17 (.28) | .16 (.27)
  Week 3 | -.28 (.89) | -.23 (.28) | .04 (.44) | .28 (.26)
  Week 4 | -.47 (.79) | -.12 (.40) | .14 (.51) | .27 (.32)
  Week 5 | -.41 (.91) | -.19 (.54) | -.01 (.38) | .42 (.43)
  Week 6 | -.69 (.93) | -.14 (.49) | -.03 (.36) | .41 (.45)

4. Secondary Outcome: Treatment Emergent Adverse Events (TEAEs) Across the Six-week Treatment Period Measure of Direct Comparison of the 4 Titration Conditions Across 6 Weeks of Treatment.
Description: Number of TEAEs across the the four titration conditions over the six-week treatment period. A score of 0 indicates no TEAEs. Higher numbers indicate greater TEAEs.
Time Frame: At the end of each week of treatment for 6 weeks.
Population: All participants who completed the protocol are included in the analysis. However, zero participants withdrew from the study after starting the study drug.
Measure: Number; unit: TEAEs
Arm/Group | Placebo | PER 1 Week Titration | PER 2 Week Titration | PER 4 mg
Number analyzed (Participants) | 2 | 3 | 6 | 8
TEAEs | 5 | 9 | 9 | 11

5. Secondary Outcome: Dropouts Across the Six-week Treatment Period Measure of Direct Comparison of the 4 Titration Conditions Across 6 Weeks of Treatment.
Description: Number dropouts across the the four titration conditions over the six-week treatment period. A score of 0 indicates no dropouts. Higher numbers indicate greater dropouts.
Time Frame: At the end of each week of treatment for 6 weeks.
Population: All participants included in analysis. However, zero participants withdrew from the study after starting the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | PER 1 Week Titration | PER 2 Week Titration | PER 4 mg
Number analyzed (Participants) | 2 | 3 | 6 | 8
Participants | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 8 weeks.
Arm/Group | Placebo | PER 1 Week Titration | PER 2 Week Titration | PER 4 mg
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/3 | 0/6 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/3 | 0/6 | 0/8
Other Adverse Events (participants affected / at risk) | 1/2 | 2/3 | 5/6 | 7/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=2) | PER 1 Week Titration (N=3) | PER 2 Week Titration (N=6) | PER 4 mg (N=8)
Cyst in Nose (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Difficulty with concentration and word finding (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Fatigue (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3) | 4 (5)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Fall (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Problems with coordination (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Balance Problems/Unsteadiness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Irritability (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lip Cramping/Twitching (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sore Throat (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fever (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hair Thinning (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Leg Abrasion (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sleep Disturbance (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypertension (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Loss of muscle definition/fat distribution (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Low White Blood Cell Count (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Low glucose level (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cognitive Change: Slowing (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Weight Gain (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
COVID-19 Infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Enrollment was delayed due to the COVID-19 pandemic. The sponsor then decided to no longer fund the study. These caused total enrollment to be low, preventing statistical analyses from being conducted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-02): https://cdn.clinicaltrials.gov/large-docs/07/NCT04417907/Prot_SAP_000.pdf